## Preoperative survey to evaluate patient allergy list, type of response to listed medication, and its relevance to perioperative care

NCT05670756

May 3, 2023

Preoperative survey to evaluate patient allergy list, type of response to listed medication, and its relevance to perioperative care - Statistical analysis

Continuous variables will be summarized using the median and interquartile ranges. Categorical variables will be presented as frequencies and percentages. Statistical analysis will be conducted using Stata (version 16; StataCorp, College Station, TX).